CLINICAL TRIAL: NCT00948311
Title: Development of an Instrument to Screen for Eating Disorder Symptoms in Persons With Type 1 Diabetes
Brief Title: Develop and Validate a Self-Administered Instrument That Will Screen for Eating Disorder Symptoms in Persons Aged 12 and Older With Type 1 Diabetes.
Status: Completed | Type: Observational
Sponsor: HealthPartners Institute (Other)
Collaborators: International Diabetes Center at Park Nicollet (Other); Park Nicollet Eating Disorder Institute (Other); Park Nicollet Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 03798-08-A
Record Dates: First submitted 2009-07-27; First posted 2009-07-29 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Type 1 Diabetes; Eating Disorder
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Feeding and Eating Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to develop and validate a survey instrument to be used by persons with type 1 diabetes aged 12 and older to screen for an eating disorder.

DETAILED DESCRIPTION:
Phase 1 - Develop an initial instrument and start to establish content validity. What do dually diagnosed patients believe are the most important, relevant, and significantly contributing constructs that we should measure in order to capture those individuals with type 1 diabetes who may exhibit symptoms of an eating disorder? What individual items will best measure these constructs?

Phase 2 - Conduct individual interviews for cognitive testing of our instrument and further examine its content validity. How well do the individual items included in our instrument capture eating disorder symptoms in patients with type 1 diabetes? Do these items accurately capture the information we seek to collect? What symptoms have we not considered? How readable and understandable are our questions?

Phase 3 - Explore the internal consistency reliability and construct validity of our instrument. Do the items in our instrument accurately capture the constructs we wish to measure? Do similar items "hang together" in a manner that is clinically and theoretically meaningful?

Phase 4 - Address convergent and discriminant validity as well as test-retest reliability. Does our instrument demonstrate appropriate convergent and divergent validity as well as test-retest reliability? Does our instrument capture eating disorder symptoms among persons with diabetes? Is our instrument more specific to the population of individuals with diabetes than traditional eating disorder instruments (i.e., does our instrument capture more information and give a more accurate presentation than the other instruments)?

ELIGIBILITY:
Inclusion Criteria:

* eating disorder
* type 1 diabetes

Exclusion Criteria:

* none

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: International Diabetes Center patient with type 1 diabetes and an eating disorder.
Sampling Method: Non-Probability Sample
Enrollment: 279 (Actual)
Dates: Start 2008-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Powers, PhD, Principal Investigator — International Diabetes Center at Park Nicollet
Locations (1):
- International Diabetes Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Papers have been published on the study.

REFERENCES:
- [Derived] Powers MA, Richter SA, Ackard DM, Craft C. Diabetes Distress Among Persons With Type 1 Diabetes. Diabetes Educ. 2017 Feb;43(1):105-113. doi: 10.1177/0145721716680888. Epub 2016 Dec 8. PMID 27932687
- [Derived] Powers MA, Richter SA, Ackard DM, Cronemeyer C. Eating disorders in persons with type 1 diabetes: A focus group investigation of early eating disorder risk. J Health Psychol. 2016 Dec;21(12):2966-2976. doi: 10.1177/1359105315589799. Epub 2015 Jun 29. PMID 26124085